CLINICAL TRIAL: NCT04554277
Title: Medico-economic Evaluation of Therapeutic Adaptation Guided by the Soluble Suppression of Tumorigenicity 2 (sST-2) Biomarker in the Management of Patients With Acute Heart Failure
Acronym: ICAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: EURO BIO Scientific (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL19_0225; 2019-A01433-54 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Biomarker; Guided therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Usual management of heart failure. The sST-2 level will be blunted.
- Biomarker guided therapy (Experimental): Guided therapy using sST-2 monitoring at the discharge from initial hospitalisation, 6, 12, 18 and 24 months of following.
  Interventions: Biological: Biomarker guided therapy

INTERVENTIONS:
Biological: Biomarker guided therapy — Guided therapy using sST-2 monitoring at the discharge from initial hospitalisation, 6, 12, 18 and 24 months of following.
  Arms: Biomarker guided therapy

SUMMARY:
Management of patients with heart Failure remains a major health concern because of the high rate of rehospitalization, mortality and induced-cost. Biomarkers could help to guide the management of patients with heart failure (HF). Soluble suppression of tumorigenicity 2 (sST2) appears as a promising biomarker. As a working hypothesis, we postulate that sST2 values monitoring could be an helpful guide for medical management in an attempt to reduce hospital readmission.

DETAILED DESCRIPTION:
Methods : ICAME is a multicentric, blinded prospective randomized controlled trial. 710 patients originated from 10 centers will be included over a period of 12 months and follow-up for 24 months. All patients have an external evaluation at 6, 12, 18 and 24 months. They were randomized into the usual treatment group (unknown sST2 level) or the interventional treatment group, for whom sST2 level was known at all external consultation and used to guide the treatment. The primary endpoint was the QALY (Quality Adjusted Life Years). The secondary endpoints were the Cost-efficacy ratio, Cost to avoid an hospitalization for heart failure, the readmission rate for any cause at 1 month and at two years, and the evolution of cardiac remodelling determined by the collagene biomarkers.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* Hospitalization for heart failure (NTproBNP(N-terminal pro-Brain Natriuretic Peptid) ≥450 pg/ml (ou BNP ≥400 pg/ml)

Exclusion criteria:

* Waiting for heart transplantation
* Scheduled valve surgery
* No fluent french
* Not able to provide informed consent
* Hemodynamic instability
* Poor outcome during the first week.
* Pregnancy
* Participating to other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Cost-utility ratio | 2 years
  Cost will be compared between guided therapy using sST-2 levels and usual group. Utility will be derived from the French EQ5D (EuroQol 5 Dimensions), measured at 24 months.
  QALY (Quality Adjusted Life Years).

SECONDARY OUTCOMES:
Cost-efficacy ratio | 2 years
  Cost to avoid an hospitalisation for heart failure
Cost of initial hospitalisation and rehospitalisation | 2 years
  Including hospitalisation, imaging and biological analysis
Number of hospitalisation for heart failure | 30 days
Number of hospitalisation for heart failure | 2 years

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Lapeyronie Hospital, Montpellier, Occitanie
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CH Béziers, Béziers
  - CHU Caen, Caen
  - CHU Grenoble, Grenoble
  - Arnaud de Villeneuve Hospital, Montpellier
  - CHU Nimes, Nîmes
  - APHP Pompidou, Paris
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse
  - CHU Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to persons who address a reasonable request to the study director and fulfil the requirements stipulated by the French CNIL (Commission National Informatic Liberty).
Supporting Information: Study Protocol
Time Frame: 24 months after randomisation